CLINICAL TRIAL: NCT02332291
Title: Connectivity Affecting the Antidepressant REsponse (The CAARE Study)
Brief Title: Connectivity Affecting the Antidepressant REsponse Study
Acronym: CAARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Warren Taylor, Professor of Psychiatry, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 141137
Record Dates: First submitted 2014-12-30; First posted 2015-01-06 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Geriatrics; Elderly; MRI; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blinded Escitalopram / Open-Label Bupropion (Active Comparator): 8 weeks of blinded escitalopram, followed by 8 weeks of open-label bupropion xl for nonremitters
  Interventions: Drug: Escitalopram; Drug: Bupropion XL
- Blinded Placebo / Open-Label Bupropion (Placebo Comparator): 8 weeks of blinded placebo, followed by 8 weeks of open-label bupropion xl for nonremitters.
  Interventions: Drug: Bupropion XL

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10-20mg daily
  Other Names: Lexapro
  Arms: Blinded Escitalopram / Open-Label Bupropion
Drug: Bupropion XL — Bupropion XL 150-450mg daily
  Other Names: Wellbutrin XL

SUMMARY:
It can be difficult to achieve remission in individuals with late-life depression (LLD) and they often require aggressive treatment. This challenge is in part due to age-related vascular changes that are common in LLD. Successful antidepressant treatment involve changes across affective, cognitive, and default mode networks. We hypothesize that in LLD, vascular disease adversely affects response to antidepressants by disrupting connectivity of these networks. The primary goal of this project is to characterize how focal vascular damage affects regional connectivity and response to antidepressants. Based on past work and pilot data, we a priori focus on the cingulum bundle and uncinate fasciculus. These key fiber bundles connect frontal, temporal, and cingulate regions involved in cognition and affective responses. Our central hypothesis is that ischemic damage to the cingulum bundle and uncinate fasciculus contributes to structural and functional connectivity deficits of those tracts. This results in a disconnection effect that alters the function of connected regions. In turn, this increases the risk of a poor response to antidepressants.

Our approach is to enroll up to 130 adults over age 60 years with a diagnosis of Major Depressive Disorder. Subjects will complete clinical evaluation, cognitive testing, and MRI/functional MRI (fMRI) sessions, including an fMRI emotional oddball task that includes attentional and affective components. Participants will be stratified by cerebral lesion severity and randomized in a 2:1 ratio to a double-blinded 8-week trial of escitalopram or matching placebo. Those who do not remit will transition to an 8-week trial of open-label bupropion, an antidepressant with a different mechanism of action. This will allow us to determine if different and distinct circuit deficits affect response to antidepressants with different mechanisms of action while also accounting for the placebo response.

DETAILED DESCRIPTION:
Individuals with late-life depression (LLD) experience high levels of disability, mortality, and poor responses to antidepressants. The MRI hallmark of 'vascular depression' in this population is significant ischemic white matter lesion (WML) severity, a finding associated with poor antidepressant outcomes. Despite observations of diffuse white matter disease in LLD, we propose in our "disconnection hypothesis" that focal damage to fiber tracts negatively affects the function of connected regions, resultantly contributing to cognitive deficits and clinical symptoms such as depression severity and negativity bias. Focal WMLs may also reduce the likelihood of an antidepressant response when the specific antidepressant used acts on neurotransmitter systems projecting through the damaged fiber tract. This implies that the effect of tract damage on clinical response may differ between drugs with different mechanism of action.

We propose that the cingulum bundle (CB) and uncinate fasciculus (UF) are key tracts in LLD as they are components of cognitive, affective and default mode networks and contain monoamine neurotransmitter projections. Supporting our model, past work implicates CB and UF deficits in LLD and our new pilot data associates tract damage with poor antidepressant response.

In a cohort of up to 130 depressed elders we will test our central hypotheses: a) focal CB and UF WMLs disrupt connectivity and function of connected regions and contribute to cognitive deficits and affective symptoms; and b) antidepressants acting on neurotransmitter systems projecting through these tracts will be less effective.

Overall Study Design: After obtaining informed consent, we will assess for eligibility. Individuals who meet eligibility criteria will complete neuropsychological testing and a one-hour magnetic resonance imaging (MRI). Subjects will then be randomized in a 2:1 ratio to receive either blinded escitalopram or identical placebo. After 8 weeks of study drug, they will be assessed for remission. Those whose depression has remitted will end their study participation. Those who remain symptomatic will be transitioned to open-label bupropion for 8 weeks, after which their participation will end. We will work with participants on plans for clinical care after the study and will offer two additional visits to facilitate that transition.

Specific Aim 1: To characterize the effect of cingulum bundle (CB) and uncinate fasciculus (UF) WMLs on tract connectivity, function of connected regions, and the cognitive and affective presentation of LLD.

Hypothesis 1: Greater CB WML volume is associated with a) reduced resting-state connectivity of frontal, temporal, and cingulate regions and b) deficits in attention, memory and processing speed.

Hypothesis 2: Greater UF WML volume is associated with a) reduced resting state functional connectivity between frontocingulate and medial temporal regions, and b) greater depression severity and negativity bias.

Exploratory Hypothesis: Greater CB WML volume is associated with failure of anterior and posterior default mode network nodes to deactivate during attentional components of the fMRI task. Greater UF WML volume is associated with greater medial temporal reactivity during the functional MRI task.

Specific Aim 2: To determine whether deficits in tract structural / functional connectivity predict nonremission to antidepressant treatments and if these relationships vary based on antidepressant mechanism of action.

Hypothesis 3: Nonremission to escitalopram will be predicted by: a) greater WML volume in the CB and UF, and b) reduced resting functional connectivity between structures connected by the CB and UF. Greater WML severity and reduced functional connectivity in these tracts will not significantly predict response to placebo.

Hypothesis 4: Nonremission to bupropion will be predicted by a) greater WML volume in the UF but not CB, and b) reduced resting functional connectivity deficits between structures connected by the UF but not CB.

Exploratory Aims: Expl. Aim 1) To determine if specific cognitive measures may serve as markers of focal tract WML damage. Expl. Aim 2) To use whole-brain multimodal imaging approaches to examine how connectivity differences in other brain regions may also predict nonremission to antidepressants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or older.
2. Current diagnosis of major depressive disorder (DSM-IV-TR), single episode, recurrent or chronic, without psychotic features, as detected by Mini-International Neuropsychiatric Inventory (MINI) and clinical exam.
3. Minimum MADRS score ≥ 15.
4. Mini-Mental State Exam ≥ 24.
5. Fluent in English.

Exclusion Criteria:

1. Current or past diagnoses of other Axis I psychiatric disorders, except for generalized anxiety disorder (GAD) symptoms occurring during a depressive episode
2. History of alcohol or drug dependence or abuse in the last three years
3. History of developmental disorder or Intelligence Quotient score < 70
4. Presence of acute suicidality
5. Acute grief (< 1 month)
6. Current or past psychosis
7. Primary neurological disorder, including but not limited to dementia, stroke, brain tumors, epilepsy, Parkinson's disease, or demyelinating diseases
8. MRI contraindications
9. Any physical or intellectual disability adversely affecting ability to complete assessments
10. Electroconvulsive therapy in last 6 months
11. Use of antidepressant medications or other psychotropic medications in the last 4 weeks (or the last 6 weeks for fluoxetine). Occasional use of benzodiazepines or non-benzodiazepine sedatives (such as zolpidem, eszopiclone, or zaleplon) during this period is allowable.
12. A failed therapeutic trial of escitalopram in the current depressive episode (defined as at least 6 weeks of treatment at a daily dose of 10mg or higher)
13. Known allergy or hypersensitivity to escitalopram or bupropion
14. Current or planned psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, MD, MHSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Ahmed R, Boyd BD, Elson D, Albert K, Begnoche P, Kang H, Landman BA, Szymkowicz SM, Andrews P, Vega J, Taylor WD. Influences of resting-state intrinsic functional brain connectivity on the antidepressant treatment response in late-life depression. Psychol Med. 2023 Oct;53(13):6261-6270. doi: 10.1017/S0033291722003579. Epub 2022 Dec 9. PMID 36482694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened in April 2015, with the first participant enrolled in June 2015. Enrollment remained open through March 2020. Recruitment involved outpatients at Vanderbilt University Medical Center, recruited through clinical referrals and community advertisements.
Pre-assignment Details: Participants enrolled while on an antidepressant medication had that medication discontinued over several weeks. At least two weeks elapsed between last antidepressant use and randomization.
  Participants enrolled at screening were excluded from the study before baseline and randomization due to a) identification of potential MRI contraindications or b) remission of depression symptoms before the baseline visit.
Groups:
- Blinded Escitalopram / Open-Label Bupropion: 8 weeks of blinded escitalopram. Remission status then assessed. If not remitting, blinded escitalopram is stopped and participants begin 8 weeks of open-label bupropion xl
  Escitalopram: Escitalopram 10-20mg daily
  Bupropion XL: Bupropion XL 150-450mg daily
- Blinded Placebo / Open-Label Bupropion: 8 weeks of blinded placebo. Remission status then assessed. If not remitting, blinded placebo is stopped and participants begin 8 weeks of open-label bupropion xl
  Placebo: 1-2 tablets daily
  Bupropion XL: Bupropion XL 150-450mg daily
Period: Phase 1: Blinded Escitalopram or Placebo
Arm/Group | Blinded Escitalopram / Open-Label Bupropion | Blinded Placebo / Open-Label Bupropion
Started | 63 | 32
Completed | 59 | 23
Not Completed | 4 | 9
Not completed — Adverse Event | 3 | 5
Not completed — Worsening Depression | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0
Period: Phase 2: Open-Label Bupropion
Arm/Group | Blinded Escitalopram / Open-Label Bupropion | Blinded Placebo / Open-Label Bupropion
Started | 22 | 19
Completed | 19 | 11
Not Completed | 3 | 8
Not completed — Adverse Event | 2 | 7
Not completed — Worsening Depression | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized in 2:1 drug:placebo ratio.
Groups:
- Blinded Placebo / Open-Label Bupropion: 8 weeks of blinded placebo. Remission status then assessed. If not remitting, blinded escitalopram is stopped and participants begin 8 weeks of open-label bupropion xl
  Placebo: 1-2 tablets daily
  Bupropion XL: Bupropion XL 150-450mg daily
- Total: Total of all reporting groups
Arm/Group | Blinded Escitalopram / Open-Label Bupropion | Blinded Placebo / Open-Label Bupropion | Total
Number analyzed (Participants) | 63 | 32 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.38 (4.86) | 66.44 (4.81) | 66.40 (4.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 20 | 56
  Male | 27 | 12 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 59 | 31 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 56 | 29 | 85
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 32 | 95
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a clinician-administered scale assessing depression severity. The range is 0-60, with higher scores representing greater depression severity
  units on a scale | 26.32 (5.00) | 25.78 (6.29) | 26.14 (5.44)
Mini-Mental State Exam (MMSE) Score [Mean (Standard Deviation); unit: units on a scale] — The MMSE is a screening questionnaire for cognitive impairment. Scores range from 0-30, with lower scores indicating poorer cognitive performance.
  units on a scale | 29.43 (0.87) | 29.22 (1.21) | 29.36 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Remission of Depression
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated measure of depression severity. Higher scores indicate greater depression severity, ranging 0-60. This will be used to define remission as a final score of 7 or less
Time Frame: From Baseline up to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Escitalopram / Open-Label Bupropion | Blinded Placebo / Open-Label Bupropion
Number analyzed (Participants) | 63 | 32
Participants | 37 | 13
Statistical Analysis 1: Comparison: Blinded Escitalopram / Open-Label Bupropion vs Blinded Placebo / Open-Label Bupropion; Statistical analyses utilized a logistic regression model with remission status (defined as final MADRS <= 7) as the dependent variable. The independent variable of interest was treatment arm assignment, and the model included age, sex, and baseline depression severity by MADRS as covariates; Test type: Superiority; p = 0.0689, Regression, Logistic — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was < 0.05; Odds Ratio, log = 0.8642, Standard Error of Mean 0.4750

2. Secondary Outcome: Change in Depression Severity, Clinician Rated
Description: Depression severity was measured by a study clinician using the MADRS. Higher scores indicate greater depression severity, ranging 0-60. Change calculated as Final MADRS - Baseline MADRS, so a negative score means greater improvement.
Time Frame: Baseline to week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Blinded Escitalopram: 8 weeks of blinded escitalopram.
  Escitalopram: Escitalopram 10-20mg daily
- Blinded Placebo: 8 weeks of blinded placebo.
  Placebo: 1-2 tablets daily
Arm/Group | Blinded Escitalopram | Blinded Placebo
Number analyzed (Participants) | 63 | 32
score on a scale | -13.90 (9.38) | -6.09 (8.90)
Statistical Analysis 1: Comparison: Blinded Escitalopram vs Blinded Placebo; Statistical analyses utilized mixed model. MADRS score was the repeated measures dependent variable. Independent variables included time, age, sex, and treatment assignment. The primary variable of interest for this analysis was an interaction term between time and treatment assignment. A statistically significant interaction term would indicate that one treatment arm experienced a greater change in MADRS score over time than the other treatment arm; Test type: Superiority; p = 0.0001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was p < 0.05; 344 degrees of freedom; Slope, fixed effect = -1.066, Standard Error of Mean 0.264

3. Secondary Outcome: Change in Depression Severity, Self Rated
Description: Self-rated depression severity was measured by the Quick Inventory of Depressive Symptoms, Self-Rated (QIDS-SR16). The QIDS-SR16 is a self-report of depression severity ranging from 0-27, with higher scores indicating greater depression severity.
Time Frame: Baseline to week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Escitalopram | Blinded Placebo
Number analyzed (Participants) | 63 | 32
units on a scale | -4.87 (5.33) | -2.09 (4.13)
Statistical Analysis 1: Comparison: Blinded Escitalopram vs Blinded Placebo; Statistical analyses utilized mixed models, with QIDS score being the repeated measures dependent variable. Independent variables included time, age, sex, and treatment assignment. The primary variable of interest was an interaction term between time and treatment assignment; Test type: Superiority; p = 0.0483, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was < 0.05; 150 degrees of freedom; Slope, fixed effects = -0.3117, Standard Error of Mean 0.1566

4. Secondary Outcome: Change in Depression Severity, Clinician Rated
Description: Change in depression severity will be measured by the MADRS. Higher scores indicate greater depression severity, ranging 0-60. Change calculated as Final MADRS - Baseline MADRS, so a negative score means greater improvement.
Time Frame: Week 8 to week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-label Bupropion XL: Bupropion XL was administered open-label for 8 weeks with flexible dosing.
  Bupropion XL: Bupropion XL 150-450mg daily
Arm/Group | Open-label Bupropion XL
Number analyzed (Participants) | 41
units on a scale | -8.75 (8.27)
Statistical Analysis 1: Comparison: Open-label Bupropion XL; Statistical analyses utilized mixed models, with MADRS score being the repeated measures dependent variable. Independent variables included time, age, and sex. The primary variable of interest was time, to indicate a change in depression severity over time with open-label treatment; Test type: Other — Analyses tested for effects of time in this one-arm, open-label study phase; p < 0.0001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was p < 0.05; 128 degrees of freedom; Slope, fixed effect = -1.186, Standard Error of Mean 0.181

5. Secondary Outcome: Change in Depression Severity, Self Rated
Description: Change in self-reported depression severity was measured by the Quick Inventory of Depressive Symptoms, Self-Rated (QIDS-SR16). This scale ranges from 0-27, with higher scores indicating greater depression severity. Change is calculated as final score less baseline score, so a negative value indicates a decrease in depression severity.
Time Frame: Week 8 to week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Bupropion XL
Number analyzed (Participants) | 41
units on a scale | -2.83 (3.85)
Statistical Analysis 1: Comparison: Open-label Bupropion XL; Statistical analyses utilized mixed models, with QIDS score being the repeated measures dependent variable. Independent variables included time, age, and sex. The primary variable of interest was time, to indicate a change in depression severity over time with open-label treatment; Test type: Other — Analyses tested for effects of time in this one-arm, open-label study phase; p = 0.0123, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was p < 0.05; 61 degrees of freedom; Slope, fixed effects = -0.2342, Standard Error of Mean 0.0908

6. Other Pre Specified Outcome: Apathy Evaluation Scale (AES)
Description: The AES is a self-report scale of apathy symptoms. The scale ranges from 18-72, with higher scores indicating greater levels of apathy. Change is calculated as final AES score - baseline AES score, so a more negative value indicates greater improvement in that symptom.
Time Frame: Baseline and Week 8
Population: Only 72 subjects out of possible 95 individuals included, as both baseline and week 8 AES data were missing for 23 participants who did not complete the self-report questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Escitalopram | Blinded Placebo
Number analyzed (Participants) | 50 | 22
units on a scale | -4.52 (7.72) | -3.00 (8.5)
Statistical Analysis 1: Comparison: Blinded Escitalopram vs Blinded Placebo; Statistical analyses used a linear model. Final AES score at week 8 was the dependent variable. Independent variables included age, sex, baseline AES score, baseline MADRS score, and treatment assignment. Treatment assignment was the independent variable of interest; Test type: Superiority; p = 0.742, Regression, Linear — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was p < 0.05; Slope = -0.636, Standard Error of Mean 1.924

7. Other Pre Specified Outcome: Ruminative Response Scale (RRS)
Description: The RRS is a self-report questionnaire assessing rumination, or responding to distress by passively focusing on the possible causes and consequences of one's distress. The RRS ranges from scores of 0-66, with higher scores indicating greater severity of rumination. Change is calculated as final RRS score - baseline RRS score, so a negative change indicates improvement in this symptom.
Time Frame: Baseline and Week 8
Population: Only 71 participants out of a possible 95 were included in analyses as either baseline or week 8 RRS data were missing for the remaining 24 participants, who did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Escitalopram | Blinded Placebo
Number analyzed (Participants) | 49 | 22
units on a scale | -10.27 (9.96) | -5.41 (10.22)
Statistical Analysis 1: Comparison: Blinded Escitalopram vs Blinded Placebo; Statistical analyses used a linear regression model. Final RRS score at week 8 was the dependent variable. Independent variables included age, sex, baseline RRS score, baseline MADRS score, and treatment assignment. Treatment assignment was the independent variable of interest; Test type: Superiority; p = 0.0232, Regression, Linear — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was p < 0.05; Slope = -5.4705, Standard Error of Mean 2.352

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during participants' duration in the study following randomization. This lasted for 8 weeks for the randomized, blinded escitalopram or placebo phase, and an additional 8 weeks for individuals progressing into the subsequent open-label bupropion phase.
Groups:
- Blinded Escitalopram: 8 weeks of blinded escitalopram
  Escitalopram: Escitalopram 10-20mg daily
- Blinded Placebo: 8 weeks of blinded placebo
  Placebo: Placebo 1-2 tablets daily
- Open-Label Bupropion: 8-weeks of open-label treatment with bupropion following initial randomization phase for individuals who did not remit to treatment with either blinded escitalopram or placebo.
  Bupropion XL: Bupropion XL 150-450mg daily
Arm/Group | Blinded Escitalopram | Blinded Placebo | Open-Label Bupropion
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/32 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/32 | 1/41
Other Adverse Events (participants affected / at risk) | 39/63 | 13/32 | 27/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Escitalopram (N=63) | Blinded Placebo (N=32) | Open-Label Bupropion (N=41)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Development of pyelonephritis requiring medical hospital admission for intravenous antibiotics.
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Gastrointestinal bleeding requiring medical hospitalization
Stroke, ischemic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Ischemic stroke, leading to medical hospitalization
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0) — Dehydration requiring hospital admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Escitalopram (N=63) | Blinded Placebo (N=32) | Open-Label Bupropion (N=41)
Irregular Heartbeat (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Subjective irregular heartbeat
Diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Minor Environmental Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — Minor injury reported not requiring medical care, such as superficial laceration
Dizziness / Lightheaded (Nervous system disorders) | 5 (5) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety / Tension (Psychiatric disorders) | 2 (2) | 1 (1) | 8 (8) — New onset or worsening anxiety
Irritability (Psychiatric disorders) | 0 (0) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Increased dreaming (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3) — Lifelike or vivid dreams
Diaphoresis (General disorders) | 2 (2) | 0 (0) | 0 (0)
Edema, peripheral (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (8) | 1 (1) | 0 (0)
Hot flashes (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 7 (7) | 0 (0) | 0 (0)
Appetite loss (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia / Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Single-site study; some missing data for self-report other outcome data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02332291/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02332291/ICF_001.pdf